CLINICAL TRIAL: NCT03197168
Title: Implementing a Psychosocial Intervention to Reduce Self-stigma and Improve Quality of Life Among Mental Health Outpatients in Chile: a Pilot Randomized Controlled Trial
Brief Title: Psychosocial Intervention to Reduce Self-stigma and Improve Quality of Life Among People With Mental Illness in Chile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Collaborators: Ministry of Health, Chile (Other Government)
Responsible Party: Principal Investigator, Franco Mascayano, BA MPH, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: SA13I20384
Record Dates: First submitted 2016-09-01; First posted 2017-06-23 (Actual); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Schizophrenia; Bipolar Disorder; Schizoaffective Disorder
Keywords: stigma; psychosocial intervention; low-and-middle income countries
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Psychotic Disorders; Social Stigma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Intervention to reduce self-stigma among people with mental illness + Usual care
  Interventions: Behavioral: Intervention to reduce self-stigma among people with mental illness
- Control (Placebo Comparator): Usual care
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Intervention to reduce self-stigma among people with mental illness — This is a 10-session group intervention (held once a week), each lasting approximately 90 minutes, taking place where the participants receive mental health treatment.
  The intervention is informed by the following key areas: (1) recovery perspective of mental health and severe mental disorders; (2) constructivist epistemology approach to learning, using cases and users' experiences; and (3) psychotherapeutic and collective narrative practices, to address internalized problems and challenges shared among the group members, respectively.
  Arms: Intervention
Behavioral: Control — Generally, each community mental health center in Chile includes two full-time psychologists, a full-time social worker and half-time occupational therapist, nurse, and psychiatrist. This team mainly offers psychiatric medication, psychotherapy, and psycho-education for users and relatives. They do not offer any specific intervention to tackle stigma among providers.
  Arms: Control

SUMMARY:
The principal objective of this pilot trial is to evaluate the effectiveness of a psychosocial intervention to reduce self-stigma and improve treatment adherence and quality of life among people with a severe mental illness who attend to Community Mental Health Centers in Chile. The intervention is based on recovery and narrative therapy and considers 10 group sessions, mainly with patients, but also integrating relatives and professionals in some of the activities.

DETAILED DESCRIPTION:
It has been shown that stigma is one of the main barriers faced by individuals with mental illness, negatively impacting their service use and continuity of treatment. Additionally, given its impact on self-esteem, personal empowerment, and social inclusion, stigma greatly affects the quality of life of this population.

Consequently, a pilot randomized controlled trial (RCT) with two arms (intervention group vs. control group) was designed and implemented. Participants were identified and recruited from two community mental health centers located in Central Chile. The intervention group, in addition to usual care, received a psychosocial intervention based on narrative therapy, recovery and psychoeducation which was specially tailored for this population by the authors.

The sample corresponds to 76 individuals with a severe mental illness (ICD-10), currently treated in the two participating Community Mental Health Centers (COSAM). The category "severe mental illness" includes patients with diagnosis of schizophrenia, schizoaffective disorder, bipolar disorder and severe depressive disorder with psychotic symptoms. Finally, those two clinics were chosen by convenience in order to facilitate the implementation of this study.

Before and after the intervention, the participants' self-stigma (Internalized Stigma of Mental Illness, ISMI), treatment adherence (weeks in treatment), and quality of life (Sevilla Quality of Life Scale) were measured. In addition, the following control variables were also evaluated, due to their influence on the principal outcomes: 1) sociodemographic information, 2) symptom presence and severity (Positive and Negative Syndrome Scale, PANSS), and 3) alcohol consumption (The Alcohol Use Disorders Identification Test, AUDIT).

ELIGIBILITY:
Inclusion Criteria:

* People with diagnosis of severe mental illness, including the following ICD-10 disorders: schizophrenia, schizoaffective disorder, bipolar disorder, severe depressive episode with psychotic symptoms.
* No longer than 5 years since the diagnosis since the first visit to a mental health clinic.

Exclusion Criteria:

* Expressing active suicidal ideation.
* Having substance abuse or dependence alone (may have psychotic symptoms but does not meet criteria for diagnoses included).
* Presenting cognitive or other sensorial impairment which is likely to preclude reliable assessment via our interview procedures

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2014-03; Primary Completion 2015-08 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Self-stigma | Baseline (month 6); First follow-up assessment (change from Baseline ISMI scores at month 10); Second follow-up assessment (change from Baseline and 1st follow-up ISMI scores at month 14)
  Internalized Stigma of Mental Illness Scale (ISMI) (Rishter et al., 2003). A Chilean version of this instrument was used during the study.

SECONDARY OUTCOMES:
Quality of Life | Baseline (month 6); First follow-up assessment (change from Baseline CSCV scores at month 10); Second follow-up assessment (change from Baseline and 1st follow-up CSCV scores at month 14)
  Seville Quality of Life Questionnaire (CSCV) (Gómez de Regil, 2016). A Chilean version of this instrument was used during the study.
Psychopathology | Baseline (month 6); First follow-up assessment (chance from Baseline PANSS scores at month 10); Second follow-up assessment (change from Baseline and 1st follow-up PANSS scores at month 14)
  Positive and Negative Syndrome Scale (PANSS). A Chilean version of this instrument was used during the study.
Treatment adherence | Baseline (month 6); First follow-up assessment (change from Treatment Adherence Baseline at month 10); Second follow-up assessment (change from Treatment Adherence Baseline and 1st follow-up at month 14)
  Adherence to medical appointments during the study. Time remaining in treatment is estimated by counting the number of days between randomization to the time of the last mental health service received. Medical records at each community mental health center are reviewed to obtain this data.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Schilling S, Bustamante JA, Sala A, Acevedo C, Tapia E, Alvarado R, Sapag JC, Yang LH, Lukens E, Mascayano F, Cid P, Tapia T. Development of an intervention to reduce self-stigma in outpatient mental health service users in Chile. Rev Fac Cien Med Univ Nac Cordoba. 2015;72(4):284-94. PMID 27107279
- See also: Related Info — https://revistas.unc.edu.ar/index.php/med/article/view/13836